CLINICAL TRIAL: NCT03273894
Title: Perioperative Management of Temperature in Children and Influence of Hypothermia on Blood Clotting in Children.
Acronym: Peritemp
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Doc.MD.Ph.D, Brno University Hospital
Other Study IDs: Temperature KDAR 2017
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2023-02

CONDITIONS: Perioperative Hypothermia
Keywords: Hypothermia, temperature management
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be tested for coagulation abnormalities - routine coagulation tests and ROTEM
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Paediatric patients undergoing surgery in general anesthesia: Paediatric patients undergoing surgery in general anesthesia with the expected duration over 30 minutes
  Interventions: Diagnostic Test: Coagulation testing

INTERVENTIONS:
Diagnostic Test: Coagulation testing — * body temperature before the intervention
  * body temperature during the intervention including the way of measuring, each 15 minutes
  * body temperature at the end of surgery, signs of the patient's heat discomfort
  * body temperature during resting time in the postanesthesia care
  * standard coagulation tests + EXTEM, FIBTEM - after anesthesia induction
  * blood sampling for standard coagulation tests (prior to the end of the surgical intervention) + EXTEM, FIBTEM.
  * if body temperature is below 34°C, two sets of ROTEM tests are run: one at patient's body temperature, following by another one at a standard temperature (37°C).
  Other Names: Coagulation status

SUMMARY:
Perioperative hypothermia carries high risk of associated complications. In the observational study, the standard perioperative temperature management will be evaluated and the influence of the hypothermia on the coagulation system according to routine coagulation testing in combination with ROTEM will be evaluated.

DETAILED DESCRIPTION:
Perioperative hypothermia is one of the complications of surgical interventions in total or regional anaesthesia. It is defined as a drop in body core temperature under 36°C. It occurs as a result of combination of anaesthesia, effecting of central thermoregulation control, environment temperature (i.e. operating theatre) and unsufficient isolation combined with patient's unability to actively warm up. As the body temperature drop in patients under anaesthesia is very frequent, body temperature checks became part of surgical patients care optimalisation. Furthermore, it is associated with complications, such as higher incidency of surgical wound infection, elongated healing process, longer time spent in a hospital, cardiac complications, elongated effect of most of anaesthetics, immunity and blood clotting disorders. Hypothermia elongates the initial phase of coagulation and results in thrombocytes malfunction. Normothermia reduces blood loss.

This prospective observative study has two parts. In the first one, investigators will evaluate the perioperative management of temperature in paediatric patients in Department of children anaesthesia and intensive care, University hospital Brno, Czech republic, where is intended to involve 1,000 patients. In the second phase, the patients who, based on the first phase of the study, would be the most prone to perioperative hypothermia, will be examined for any change of coagulation parameters related to the hypothermia. Investigators intend to involve 100 consecutive patients of the original group. The examined parameters are standard coagulation tests, EXTEM, FIBTEM tests obtained from a rotational thromboelastometry, or other ROTEM test related to the particular pathology. Investigators will use a standardized method of fluid management to affect dilutional coagulopathy.

Standard perioperative patient's monitoring - temperature sensor monitoring of body temperature, ECG, noninvasive blood pressure, oxygen saturation, EtCO2

Temperature management:

- the anaesthetist decides if some warming tools are needed and notes the used ones, which involve: warmed infusion, heating blanked, air warming system, infusion pipe heater, increasing of temperature in the operating theatre, covering the patient or another method of temperature management

Monitored parameters in the first phase:

* body temperature before the intervention (measured in the office previously), operating theatre's temperature at the beginning of anaesthesia
* body temperature during the intervention including the way of measuring, marked each 15 minutes
* body temperature at the end of the entire intervention, including signs of the patient's heat discomfort
* body temperature during resting time in the after-surgery resting room

Monitored parameters in the second phase:

* monitored parameters in the first phase + following:
* blood sampling for standard coagulation tests (following initial of general anaesthesia) + EXTEM, FIBTEM. In case of any pathology found here, more relevant test are run. The test is analysed by anaesthetist or ICU doctor, where the ROTEM machine is.
* blood sampling for standard coagulation tests (prior to the end of the surgical intervention) + EXTEM, FIBTEM. In case of any pathology found here, more relevant test are run. The test is analysed by anaesthetist or ICU doctor, where the ROTEM machine is.
* if body temperature is below 34°C, two sets of ROTEM tests are run: one at patient's body temperature, following by another one at a standard temperature (37°C).

Statistic evaluation:

* demographic - age, sex, type of surgery, duration of surgery, type of anaesthesia
* changes of core temperature during the perioperative care and influence of used warming tools, side effects of changes of core temperature
* laboratory tests - standard coagulation tests and ROTEM - EXTEM, FIBTEM test

ELIGIBILITY:
Inclusion Criteria:

* paediatric patients of age 0 - 18 years (+ 364 days) indicated to a surgical intervention with expected duration longer than 30 minutes
* informed consent of the patient's legal representative to blood sampling in order to run the coagulation tests

Exclusion Criteria:

* surgical intervention shorter than 20 minutes for the second phase:
* disagreement of the patient and their legal representative
* preexisting blood clotting disorder
* potential damage on the patient caused by non-indicated blood sampling (newborns with low, very low or extremely low birth weight)

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric patients undergoing surgery in general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Influence of the hypothermia on the coagulation status | Perioperatively
  Perioperative temperature management will be evaluated and the blood samples will be tested for possible coagulation abnormalities in patients undergoing surgery in general anesthesia

SECONDARY OUTCOMES:
Temperature management | Perioperatively
  Data will be evaluated and each perioperative temperature management method will be validated for the effectivity

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, prof.MD.Ph.D, Study Chair — Brno University Hospital
Locations (1):
- University hospital Brno, Brno, Jihomoravská Kraj, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Trckova A, Bonischova T, Zelinkova H, Stourac P. Perioperative temperature management and coagulation: effects of mild hypothermia in a prospective study. Front Med (Lausanne). 2025 Jun 16;12:1536782. doi: 10.3389/fmed.2025.1536782. eCollection 2025. PMID 40589964